CLINICAL TRIAL: NCT03734146
Title: Independent and Combined Effects of Aerobic and Resistance Training on Blood Pressure
Acronym: ART-B
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Iowa State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 14-330
Record Dates: First submitted 2018-10-31; First posted 2018-11-07 (Actual); Last update posted 2018-11-07 (Actual); Status verified 2018-10

CONDITIONS: Cardiovascular Risk Factor
MeSH Terms: interventions — Exercise; Resistance Training

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor was blinded to treatment group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Aerobic exercise (AE) (Experimental): Engage in supervised aerobic exercise for 60 minutes on 3 days per week for 8 weeks. Exercise is performed on a recumbent bike or treadmill at 50-80% of their heart rate reserve.
  Interventions: Behavioral: Aerobic Exercise
- Resistance exercise (RE) (Experimental): Engage in supervised resistance exercise for 60 minutes on 3 days per week for 8 weeks. Exercise consists of 3 sets of 8-12 repetitions of 12 exercises for the major muscle groups.
  Interventions: Behavioral: Resistance Exercise
- Combined Resistance and Aerobic Exercise (Experimental): Engage in supervised aerobic resistance exercise for 60 minutes on 3 days per week for 8 weeks. Exercise consists of 30 min aerobic exercise at 50-80% heart rate reserve and 30 min of resistance exercise comprising 2 sets of 8-12 repetitions of 9 exercises for the major muscle groups.
  Interventions: Behavioral: Combined aerobic and resistance exercise
- No training control (No Intervention): No exercise training. Participants will refrain from any moderate-vigorous exercise or resistance training for 8 weeks.

INTERVENTIONS:
Behavioral: Aerobic Exercise — 180 minutes of moderate-vigorous intensity aerobic exercise per week
  Arms: Aerobic exercise (AE)
Behavioral: Resistance Exercise — 180 minutes of resistance exercise per week
  Arms: Resistance exercise (RE)
Behavioral: Combined aerobic and resistance exercise — 180 minutes of exercise per week with 90 minutes per week coming from moderate-vigorous intensity aerobic exercise and 90 minutes per week coming from resistance exercise
  Arms: Combined Resistance and Aerobic Exercise

SUMMARY:
We compared the effects of 8 weeks of aerobic exercise only, resistance exercise only, or a combination of both on blood pressure in overweight or obese middle-aged adults with elevated blood pressure. Participants engaged in supervised exercise sessions 3 times per week for 60 minutes each session. Outcomes were assessed at baseline and after the 8-week intervention. Extra-intervention physical activity and diet were also assessed.

ELIGIBILITY:
Inclusion Criteria:

* Systolic/diastolic blood pressure of 120-159/80-99 mm Hg
* Non-smoking
* Overweight or obese, with a body mass index of 25-40 kg/m2
* Inactive--not meeting the aerobic or resistance physical activity guidelines, which means engaging in less than 150 minutes/wk of moderate intensity aerobic exercise and less than 2 days per week of resistance training over the past 3 months.

Exclusion Criteria:

* Unstable coronary heart disease or decompensated heart failure
* Severe pulmonary hypertension or aortic stenosis
* Acute myocarditis, endocarditis, pericarditis, or aortic dissection
* Other medical condition that is life-threatening or that can interfere or be aggravated by the exercise training such as cancer, uncontrolled diabetes, severe pain or mobility limitations.
* Premenopausal women or postmenopausal women taking hormonal replacement therapy
* Pregnant women or anticipated pregnancy via IVF or other medical procedures during the course of the intervention

Ages: 45 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2014-07-15 (Actual); Primary Completion 2014-12-19 (Actual); Study Completion 2014-12-19 (Actual)

PRIMARY OUTCOMES:
Change in resting blood pressure | Immediately before and after the 8 week intervention
  resting systolic and diastolic blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Duck-chul Lee, PhD, Principal Investigator — Iowa State University

IPD SHARING:
Plan to Share IPD: No